CLINICAL TRIAL: NCT04217330
Title: HomeBase2: An Implementation Trial to Improve Access to Pulmonary Rehabilitation in People With Chronic Obstructive Pulmonary Disease
Brief Title: An Implementation Trial to Improve Access to Pulmonary Rehabilitation in People With COPD
Acronym: HomeBase2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Institute for Breathing and Sleep, Australia (Other); University of Melbourne (Other); La Trobe University (Other); Thoracic Society of Australia and New Zealand (Unknown); Lung Foundation Australia (Unknown)
Responsible Party: Principal Investigator, Anne E Holland PhD, FThorSoc, Professor of Physiotherapy, Monash University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55803
Record Dates: First submitted 2019-12-17; First posted 2020-01-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary rehabilitation; Implementation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be informed that the trial is assessing the impact of pulmonary rehabilitation models on patient and health system outcomes, but not the specific nature of the models of interest, or the intervention group to which their site has been allocated.
  Assessors will be blinded to the site allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Pulmonary rehabilitation programs assigned to the intervention group will offer eligible participants the choice of participating in an 8-week program of either home-based pulmonary rehabilitation or traditional centre-based pulmonary rehabilitation.
  Interventions: Behavioral: Choice of home-based or centre-based pulmonary rehabilitation
- Control (Active Comparator): Pulmonary rehabilitation programs assigned to the control group will offer eligible participants the opportunity to participate in an 8-week centre-based pulmonary rehabilitation program, as per current practice.
  Interventions: Behavioral: Centre-based pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Choice of home-based or centre-based pulmonary rehabilitation — Participants will be offered the choice of HomeBase, a home-based pulmonary rehabilitation program, or the traditional centre-based pulmonary rehabilitation program.
  Arms: Intervention
Behavioral: Centre-based pulmonary rehabilitation — Participants will be offered a traditional centre-based pulmonary rehabilitation program
  Arms: Control

SUMMARY:
People with chronic obstructive pulmonary disease (COPD) experience distressing breathlessness and high health care utilisation. There is compelling evidence that pulmonary rehabilitation improves symptoms and reduces hospitalisation, but is delivered to <10% of patients who would benefit. The investigators developed a low cost model of pulmonary rehabilitation that can be delivered entirely at home. The HomeBase model had equivalent outcomes to centre-based pulmonary rehabilitation in a phase II efficacy trial, with higher completion rates. The investigators hypothesise that a patient centred model offering a choice between home or centre-based pulmonary rehabilitation may increase program completion rates, with improved outcomes for patients and the health system.

This is a cluster randomised implementation trial investigating whether offering a choice of home or centre-based pulmonary rehabilitation can reduce hospitalisation, improve pulmonary rehabilitation completion and enhance patient outcomes in people with COPD. 14 pulmonary rehabilitation programs located across Australia will each recruit 35 people with COPD. Intervention centres: People with COPD will be offered the choice of centre-based pulmonary rehabilitation or the HomeBase model. Comparison centres: Only the existing centre-based model will be offered. The primary outcome is all cause, non-elective hospitalisation at 12 months. Other outcomes are symptoms, exercise capacity and quality of life at 8 weeks and 12 months; and health care costs at 12 months for full economic evaluation.

ELIGIBILITY:
Inclusion criteria for pulmonary rehabilitation programs:

• Outpatient pulmonary rehabilitation programs that admit at least 50 people with COPD each year.

Inclusion criteria for participants:

* Diagnosis of COPD confirmed on spirometry
* Able to read, write and speak English
* Able to provide informed consent.

Exclusion Criteria:

* Attended pulmonary rehabilitation within 1 year
* Comorbidities which preclude exercise training.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
All cause, non-elective hospitalisation | 12 months after completing pulmonary rehabilitation
  The number of participants hospitalised at least once will be compared between groups

SECONDARY OUTCOMES:
Change in 6-minute walk distance | End of rehabilitation and 12 months later
  Distance walked in 6 minutes
Change in chronic respiratory disease questionnaire total and domain scores | End of rehabilitation and 12 months later
  Disease-specific health-related quality of life measure; scores range 1-7, higher scores indicate better health-related quality of life
EQ-5D-5L | End of rehabilitation and 12 months later
  Generic health-related quality of life measure to inform economic analysis; 5 dimensions each scored 1-5 with lower values indicating better health-related quality of life
Change in dyspnoea-12 | End of rehabilitation and 12 months later
  Global measure of breathlessness; total scores range from 0 to 36, with higher scores corresponding to greater severity of dyspnoea
Change in objectively measured physical activity | End of rehabilitation and 12 months later
  Objective measure of physical activity using the actigraph
Health care costs | 12 months following pulmonary rehabilitation completion
  Health care costs in Australian dollars will be calculated using health care utilisation data including hospitalisation, primary care visits and medication use
Program completion | End of rehabilitation
  The number of participants who complete their allocated rehabilitation program (attend at least 70% of planned sessions).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Holland, Principal Investigator — Monash University
Locations (11):
- Australia (11):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Mount Druitt Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Top End Health Service, Darwin, Northern Territory
  - Prince Charles Hospital, Brisbane, Queensland
  - Central Adelaide Local Health Network, Adelaide, South Australia
  - Southern Adelaide Local Health Network, Adelaide, South Australia
  - Peninsula Health, Melbourne, Victoria
  - St John of God Frankston Rehabilitation, Melbourne, Victoria
  - Western Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make individual participant data available to other researchers for related projects with appropriate ethical oversight. The data provided would be in re-identifiable form with no identifying information provided. Access will only be granted to researchers who agree to preserve the confidentiality of the information. Access will require approval from the research team as well as approval from a Human Research Ethics Committee.
Supporting Information: Study Protocol, ICF
Time Frame: After publication of the main trial results, for 7 years.
Access Criteria: Access will only be granted to researchers who agree to preserve the confidentiality of the information. Access will require approval from the research team as well as approval from a Human Research Ethics Committee

REFERENCES:
- [Derived] Cox NS, Holland AE, Jones AW, McDonald CF, O'Halloran P, Mahal A, Hepworth G, Lannin NA. Implementation of offering choice of pulmonary rehabilitation location to people with COPD: a protocol for the process evaluation of a cluster randomised controlled trial. Trials. 2023 Mar 8;24(1):173. doi: 10.1186/s13063-023-07179-2. PMID 36890526
- [Derived] Holland AE, Jones AW, Mahal A, Lannin NA, Cox N, Hepworth G, O'Halloran P, McDonald CF. Implementing a choice of pulmonary rehabilitation models in chronic obstructive pulmonary disease (HomeBase2 trial): protocol for a cluster randomised controlled trial. BMJ Open. 2022 Apr 11;12(4):e057311. doi: 10.1136/bmjopen-2021-057311. PMID 35410931